CLINICAL TRIAL: NCT00329264
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study of the Efficacy and Safety of Sustained-Release Quetiapine Fumarate (SEROQUEL®) Compared With Placebo in the Treatment of Generalized Anxiety Disorder
Brief Title: Safety & Efficacy Study of Quetiapine Fumarate (SEROQUEL®) vs. Placebo in Generalized Anxiety Disorder
Acronym: TITANIUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00009; Titanium
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: GAD; anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate

SUMMARY:
The purpose of this study is to demonstrate that quetiapine SR (SEROQUEL®) is efficacious and safe in the acute treatment of patients with Generalized Anxiety Disorder.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented clinical diagnosis of Generalized Anxiety Disorder.
* Be able to understand and comply with the requirements of the study.
* Able to understand and provide written informed consent

Exclusion Criteria:

* Patients (female) must not be pregnant or lactating
* Current or past diagnosis of stroke or transient ischemic attack (TIA).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2006-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from randomization in the HAM-A total score at Day 57

SECONDARY OUTCOMES:
Change from randomization in CGI-S score at Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, MD, Study Director — AstraZeneca
Locations (58):
- United States (58):
  - Research Site, Springdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Encino, California
  - Research Site, Newport Beach, California
  - Research Site, Oceanside, California
  - Research Site, Redlands, California
  - Research Site, Santa Ana, California
  - Research Site, Denver, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Walton Beach, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Topeka, Kansas
  - Research Site, New Orleans, Louisiana
  - Research SIte, Fall River, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Ridgeland, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Clementon, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Friendswood, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Woodstock, Vermont
  - Research Site, Herndon, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Seattle, Washington
  - Research Site, Charleston, West Virginia

REFERENCES:
- [Derived] Montgomery SA, Locklear JC, Svedsater H, Eriksson H. Efficacy of once-daily extended release quetiapine fumarate in patients with different levels of severity of generalized anxiety disorder. Int Clin Psychopharmacol. 2014 Sep;29(5):252-62. doi: 10.1097/YIC.0000000000000026. PMID 24394383
- [Derived] Stein DJ, Bandelow B, Merideth C, Olausson B, Szamosi J, Eriksson H. Efficacy and tolerability of extended release quetiapine fumarate (quetiapine XR) monotherapy in patients with generalised anxiety disorder: an analysis of pooled data from three 8-week placebo-controlled studies. Hum Psychopharmacol. 2011 Dec;26(8):614-28. doi: 10.1002/hup.1256. Epub 2011 Dec 6. PMID 22143997
- [Derived] Khan A, Joyce M, Atkinson S, Eggens I, Baldytcheva I, Eriksson H. A randomized, double-blind study of once-daily extended release quetiapine fumarate (quetiapine XR) monotherapy in patients with generalized anxiety disorder. J Clin Psychopharmacol. 2011 Aug;31(4):418-28. doi: 10.1097/JCP.0b013e318224864d. PMID 21694613